CLINICAL TRIAL: NCT00342342
Title: Family Studies of Ocular Traits
Brief Title: Family Studies of Eye Traits
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903067; 03-HG-N067
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Cataracts; Glaucoma; Myopia
Keywords: Association; Linkage Study; Familial Aggregation; Linkage Disequilibrium
MeSH Terms: conditions — Cataract; Glaucoma; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Beaver Dam Eye Study: Individuals over 45 years of age enrolled in Beaver Dam Wisconsin
- Framingham Eye Study: Subset of individuals from the Framingham Heart Study who received eye examinations

SUMMARY:
This study will examine blood specimens from patients with various eye disorders who previously participated in the Beaver Dam Eye Study to try to identify genes responsible for these disorders. The Beaver Dam study was designed to determine the incidence and causes of age-related eye conditions, including cataract (changes in the lens of the eye that can impair vision); retinopathy (diseases of the retina - the thin layer of tissue that lines the back of the eye); age-related maculopathy (degeneration or atrophy of the macula - the center part of the retina responsible for fine vision); and impaired vision. Findings from this study and others have shown that age-related eye disorders often run in families, indicating a genetic component in their development.

All participants in the Beaver Dam study who had family members in the study may be included in the current NHGRI study. The Beaver Dam study included residents of the township of Beaver Dam, Wisconsin, who were between 45 and 84 years of age at enrollment. Participants had thorough eye examinations and blood samples drawn at baseline and 5 and 10 years after the baseline evaluation. Fifteen-year follow-ups will start in 2003.

This study will analyze data and blood samples previously collected from Beaver Dam study participants to identify genes related to numerous age-related visual traits. No new participants will be recruited.

DETAILED DESCRIPTION:
The Beaver Dam Eye Study was designed to determine the long-term incidence and causes of cataract, age-related maculopathy (ARM), retinopathy, and impaired vision. Age-related macular degeneration and cataract are leading causes of loss of vision in the United States. In Beaver Dam, preliminary analyses indicate that in those people who were 75+ years of age at the baseline examination, 72% developed nuclear cataract, 39% developed cortical cataract, 22% developed posterior subcapsular cataract (PSC); 37% developed early ARM (large soft indistinct drusen, retinal pigment epithelial (RPE) depigmentation, and increased retinal pigment); 10% developed signs of late ARM (exudative macular degeneration and geographic atrophy); 37% developed some impairment of vision; and 6% developed severely impaired vision by the 10-year follow-up. Thus, these are common problems in older persons. Because people 75 years of age and older are the most rapidly growing segment of the population with an estimated increase of over 60% in the next 25 years, these problems pose a societal burden due to the large number of older persons they will affect. Additionally, we have observed substantial familial aggregation for several of these traits: ARM, nuclear cataract, cortical cataract and ocular refraction. The primary goal of this proposal is to perform linkage analysis on data collected as part of the Beaver Dam eye study. NHGRI investigators will be involved in the analysis of coded data only. Dr. Bailey-Wilson may provide financial support to help cover the cost of DNA extraction from her budgets but NO samples will be sent to NHGRI. All NHGRI effort on this study will be funded through Dr. Bailey-Wilson s intramural budget.

In addition to the data from the Beaver Dam Eye study, we will also analyze previously existing data on glaucoma, intraocular pressure and cup-disc ratio from the Framingham Eye Study (FES) which is a substudy of the well known cohort study called the Framingham Heart Study (FHS). We will perform both linkage and association analysis of these data for comparison to the results found in the BDES data.

ELIGIBILITY:
* INCLUSION CRITERIA:

All individuals aged 45-84 years of age living in the township of Beaver Dam Wisconsin were invited to participate.

In the Framingham, cohort study, inclusion criteria were that the participants were residents of Framingham, MA or offspring of the original enrolless into the FHS.

EXCLUSION CRITERIA:

None other than not meeting the Inclusion Criteria.

In the Framingham Eye Study, enrollees from the FHS who were deceased at the time of the FES exams (1970's) would not be able to enroll.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Beaver Dam Eye study used a community sample.@@@Framingham Eye study used a subset of a community sample.
Sampling Method: Non-Probability Sample
Enrollment: 7370 (Actual)
Dates: Start 2002-12-04 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Refractive error | At study enrollment
  ocular refractive error was measured on both eyes at enrollment in both the BDES and FES

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bailey-Wilson, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (5):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland
  - Boston University, Boston, Massachusetts
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Tielsch JM, Sommer A, Witt K, Katz J, Royall RM. Blindness and visual impairment in an American urban population. The Baltimore Eye Survey. Arch Ophthalmol. 1990 Feb;108(2):286-90. doi: 10.1001/archopht.1990.01070040138048. PMID 2271016
- [Background] Klein R, Wang Q, Klein BE, Moss SE, Meuer SM. The relationship of age-related maculopathy, cataract, and glaucoma to visual acuity. Invest Ophthalmol Vis Sci. 1995 Jan;36(1):182-91. PMID 7822146
- [Background] Hiller R, Sperduto RD, Ederer F. Epidemiologic associations with nuclear, cortical, and posterior subcapsular cataracts. Am J Epidemiol. 1986 Dec;124(6):916-25. doi: 10.1093/oxfordjournals.aje.a114481. PMID 3776974